CLINICAL TRIAL: NCT03573336
Title: A Randomized, Double-blind, Parallel-group, Multicenter Phase 2b Study to Assess the Efficacy and Safety of Two Different Doses of Vilaprisan (BAY1002670) Versus Placebo in Women With Symptomatic Endometriosis
Brief Title: Assess Safety and Efficacy of Vilaprisan in Subjects With Endometriosis
Acronym: VILLENDO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15792; 2013-004768-72 (EudraCT Number)
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vilaprisan (BAY1002670) 2 mg (Experimental): Premenopausal women 18 years and older with endometriosis with randomized ratio = 1:1:1 Vilaprisan: 2 mg
  Interventions: Drug: Vilaprisan (BAY1002670)
- Vilaprisan (BAY1002670) 4 mg (Experimental): Premenopausal women 18 years and older with endometriosis with randomized ratio = 1:1:1 Vilaprisan: 4 mg
  Interventions: Drug: Vilaprisan (BAY1002670)
- Placebo group (Placebo Comparator): Premenopausal women 18 years and older with endometriosis with randomized ratio = 1:1:1
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — Intake orally, once daily
  Arms: Vilaprisan (BAY1002670) 2 mg; Vilaprisan (BAY1002670) 4 mg
Drug: Matching Placebo — Intake orally, once daily
  Arms: Placebo group

SUMMARY:
The primary objective of this study was to assess the efficacy and safety of two doses of vilaprisan compared to placebo in women with symptomatic endometriosis.

The secondary objective of this study was to evaluate the safety and tolerability of two different doses of vilaprisan in women with symptomatic endometriosis.

With the implementation of protocol version 4.0 dated 11-Dec-2018, no new subjects were enrolled. The objectives above cannot be reached as only limited data is available from subjects recruited before the temporary pause.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Pre-menopausal women 18 years (inclusive) and above at the time of Visit 1
* Women with endometriosis confirmed by laparoscopy or laparotomy OR diagnosed based on imaging
* Moderate to severe endometriosis-associated pelvic pain (EAPP)
* Adherence to screening period diary entries
* Willingness to use only standardized pain medication if needed
* Good general health (except for findings related to endometriosis)
* Normal or clinically insignificant cervical cytology not requiring further follow-up
* An endometrial biopsy performed at the screening phase without significant histological disorder
* Use of an acceptable non-hormonal method of contraception
* Willingness / ability to comply with electronic diary entry for the duration of study participation

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before Visit 1)
* Hypersensitivity to any ingredient of the study treatments
* Laboratory values outside the inclusion range before randomization, and considered clinically relevant
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug including elevated liver enzymes
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding
* Abuse of alcohol, drugs, or medicines (e.g. laxatives) as evaluated by the investigator
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results
* Endometriosis-specific treatments for symptom relief except rescue pain medication according to protocol
* Simultaneous participation in another clinical trial with investigational medicinal product(s). Participation in another trial prior to study entry that might have an impact on the study objectives, at the discretion of the investigator
* Inability to cooperate with the study procedures for any reason
* Previous assignment to treatment (e.g. randomization) during this study (allowing previously randomized subjects to be re-included into the study may lead to bias)
* Hypersensitivity to any ingredient of standardized pain medication
* Wish for pregnancy during the study
* Regular use of pain medication due to other underlying diseases
* Non-responsiveness of EAPP to GnRH-a (Gonadotropin-releasing hormone agonists)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (23):
- United States (6):
  - Office of Dr. James A. Simon, MD, Washington D.C., District of Columbia
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Southern Clinical Research Associates LLC, Metairie, Louisiana
  - Unified Women's Clinical Research - Morehead City, Morehead City, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
- Austria (4):
  - Medizinische Universität Graz, Graz, Styria
  - Kepler Universitätsklinikum Campus IV, Linz, Upper Austria
  - Universitätsklinikum AKH Wien, Vienna
  - KABEG Landeskrankenhaus Villach, Villach
- Canada (3):
  - Queen's University, Kingston, Ontario
  - Ottawa Hospital-Riverside Campus, Ottawa, Ontario
  - Clinique OVO, Montreal, Quebec
- Czechia (2):
  - Gynekologie MEDA s.r.o., Brno
  - GynCare MUDr. Michael Svec s.r.o., Pilsen
- Finland (2):
  - VL-Medi Oy, Helsinki
  - Satakunnan keskussairaala, Pori
- A.O.U.I. Verona, Verona, Veneto, Italy
- Japan (4):
  - Tokeidai Memorial Clinic, Sapporo, Hokkaido
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Toyama Prefectural Central Hospital, Toyama
- Centrum Medyczne Chodzki, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Taylor HS, Dong L, Haikonen J, Oppelt P, Tamussino K, Wenzl R, Faustmann T, Groettrup-Wolfers E, Ren X, Seitz C. Vilaprisan for the treatment of symptomatic endometriosis: results from a terminated phase 2b randomized controlled trial. F S Rep. 2024 Mar 11;5(2):189-196. doi: 10.1016/j.xfre.2024.03.002. eCollection 2024 Jun. PMID 38983729
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 7 study centers worldwide, between 04-Jul-2018 (first participant first visit) and 26-Nov-2020 (last participant last visit).
Pre-assignment Details: With the implementation of protocol version 4.0 dated 11-Dec-2018, no new participants were enrolled. The objectives of this study cannot be reached as only limited data is available from participants recruited before the treatment stopped. Overall, 48 participants were screened, of whom 8 participants were randomized and received the study treatment.
Groups:
- Vilaprisan (BAY1002670) 2 mg: Premenopausal women 18 years and older with endometriosis received the treatment of Vilaprisan 2 mg.
- Vilaprisan (BAY1002670) 4 mg: Premenopausal women 18 years and older with endometriosis received the treatment of Vilaprisan 4 mg
- Placebo: Premenopausal women 18 years and older with endometriosis received placebo.
Period: Overall Study
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Started | 2 | 4 | 2
Treated | 2 | 4 | 2
Completed | 0 | 0 | 0
Not Completed | 2 | 4 | 2
Not completed — Study terminated | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 2 | 8
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 4 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Worst Pelvic Pain (Measured on a Numerical Rating Scale [NRS], Recorded in the Daily Endometriosis Symptom Diary [ESD])
Description: Pain intensity was assessed on 11-point (0-10) NRS by ESD item 1. In ESD item 1, participants were asked to rate the worst pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. Mean 'worst pelvic pain' was calculated as the sum of the participant's daily assessments of the ESD item 1 ("worst pain" during the last 24 hours) during a study period divided by number of days with pain assessment in that study period. This was summarized by study period. No inferential statistical analysis was performed.
Time Frame: Screening period (up to a maximum of 75 days) + treatment period (up to a maximum of 168 days)
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Scores on a scale
  Screening period | 6.0 [5.3 to 6.8] | 5.8 [4.0 to 7.1] | 5.6 [5.5 to 5.7]
  Treatment period | 3.0 [2.0 to 4.0] | 3.8 [1.9 to 5.6] | 5.0 [4.1 to 5.9]

2. Secondary Outcome: Mean Worst Pelvic Pain (Measured on a Numerical Rating Scale [NRS], Recorded in the Daily Endometriosis Symptom Diary [ESD]) on Days With/Without Vaginal Bleeding
Description: Pain intensity was assessed on 11-point (0-10) NRS by ESD item 1. In ESD item 1, participants were asked to rate the worst pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. Mean 'worst pelvic pain' on bleeding/non-bleeding days was calculated as the sum of the participant's daily assessments of the ESD item 1 ("worst pain" during the last 24 hours) on bleedings/non-bleeding days during a study period divided by number of bleeding/non-bleeding days with pain assessment in that study period. This was summarized by study period. No inferential statistical analysis was performed.
Time Frame: Screening period (up to a maximum of 75 days) + treatment period (up to a maximum of 168 days)
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Scores on a scale
  Screening period: Worst Pain on days with vaginal bleeding | 6.5 [4.6 to 8.4] | 6.9 [4.9 to 8.4] | 7.0 [6.9 to 7.0]
  Screening period: Worst Pain on days without vaginal bleeding | 5.9 [5.5 to 6.3] | 5.5 [3.7 to 6.7] | 5.3 [5.1 to 5.6]
  Treatment period: Worst Pain on days with vaginal bleeding | NA [NA to NA] — No participant had pain on vaginal bleeding days in the treatment period. | 5.4 [3.8 to 7.0] | 6.0 [5.1 to 6.9]
  Treatment period: Worst Pain on days without vaginal bleeding | 3.0 [2.0 to 4.0] | 3.7 [1.8 to 5.6] | 4.7 [4.0 to 5.5]

3. Secondary Outcome: Mean Number of Tablets of Rescue Pain Medication 1 (Ibuprofen 200 mg) Taken Daily for Endometriosis-associated Pelvic Pain (EAPP)
Description: Mean number of tablets of rescue pain medication 1 (Ibuprofen 200 mg) taken daily for EAPP was calculated as the sum of the tablets taken for EAPP during a study period divided by the number of days in that study period. This was summarized by study period. No inferential statistical analysis was performed.
Time Frame: Screening period (up to a maximum of 75 days) + treatment period (up to a maximum of 168 days)
Measure: Mean (Full Range); unit: Tablets
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Tablets
  Screening period | 0.61 [0.35 to 0.86] | 1.01 [0 to 2.14] | 1.03 [0.31 to 1.74]
  Treatment period | 0.09 [0.01 to 0.17] | 0.16 [0.05 to 0.42] | 0.81 [0.33 to 1.30]

4. Secondary Outcome: Mean Number of Tablets of Rescue Pain Medication 2 (Tramadol 50 mg) Taken Daily for Endometriosis-associated Pelvic Pain (EAPP)
Description: Mean number of tablets of rescue pain medication 2 (Tramadol 50 mg) taken daily for EAPP was calculated as the sum of the tablets taken for EAPP during a study period divided by the number of days in that study period. This was summarized by study period. No inferential statistical analysis was performed.
Time Frame: Screening period (up to a maximum of 75 days) + treatment period (up to a maximum of 168 days)
Measure: Mean (Full Range); unit: Tablets
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Tablets
  Screening period | 0 [0 to 0] | 0 [0 to 0] | 0.17 [0 to 0.34]
  Treatment period | 0.01 [0 to 0.03] | 0.01 [0 to 0.05] | 0.02 [0.01 to 0.02]

5. Secondary Outcome: The Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study. TEAE is defined as AE that is observed or reported after the first administration of study drug or if it starts before the first administration of study drug and the intensity/grade worsens on treatment) in this study.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants
  Non-serious TEAEs | 2 | 3 | 2
  SAEs | 1 | 3 | 0
  Deaths | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinical Significant Abnormal Endometrial Histology Findings
Description: Number of participants with endometrial histology findings, e.g. hyperplasia, malignant neoplasm or endometrial polyps
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants
  Endometrial hyperplasia | 0 | 0 | 0
  Malignant neoplasm | 0 | 0 | 0
  Endometrial polyps | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinical Significant Abnormal Ultrasound Examinations
Description: Ultrasound examinations (evaluated for efficacy and safety) will be performed by a qualified expert in performing gynecologic ultrasound exams. If possible, the same examiner should conduct all examinations of a subject throughout the study and the same ultrasound machine (per site) should be used throughout the study. Preferably the safety evaluation should be performed by transvaginal ultrasound (TVU). However, if deemed appropriate, transabdominal or transrectal ultrasound examinations can be performed instead. The chosen method should be used consistently throughout the study.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinical Significant Abnormal Bone Mineral Density Measurements
Description: A Dual-energy X-ray absorptiometry (DEXA) scan of the lumbar spine (lumbar anterior-posterior, L1-L4) and the hip/femoral neck were performed.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Significant Abnormal Laboratory Values
Description: Clinical laboratory values including the values of hematology, general chemistry, urinalysis, coagulation, hormones, immunology and vitamins.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 2
Participants | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from first study medication intake until last visit of the subject (516 days on average).
Arm/Group | Placebo | Vilaprisan (BAY1002670) 2 mg | Vilaprisan (BAY1002670) 4 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 3/4
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Vilaprisan (BAY1002670) 2 mg (N=2) | Vilaprisan (BAY1002670) 4 mg (N=4)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Vilaprisan (BAY1002670) 2 mg (N=2) | Vilaprisan (BAY1002670) 4 mg (N=4)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bone density decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (20) | 1 (6) | 2 (27)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
No inferential statistical analysis was performed due to a small population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03573336/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03573336/SAP_000.pdf